CLINICAL TRIAL: NCT02378376
Title: In Vivo Quantification of Short Chain Fatty Acids Production in the Human Colon After Consumption of Different Cereal Fractions.
Brief Title: In Vivo Quantification of Short Chain Fatty Acids Production in the Human Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: s55383
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Wheat derived fiber fraction 1 (Experimental): Arabinoxylan oligosaccharides
  Interventions: Dietary Supplement: Arabinoxylan oligosaccharides
- Wheat derived fiber fraction 2 (Experimental): Dietary fiber enriched bran
  Interventions: Dietary Supplement: Dietary fiber enriched bran

INTERVENTIONS:
Dietary Supplement: Arabinoxylan oligosaccharides
  Arms: Wheat derived fiber fraction 1
Dietary Supplement: Dietary fiber enriched bran
  Arms: Wheat derived fiber fraction 2

SUMMARY:
During this project the amount of SCFA produced in the colon after consumption of 2 different 13C-labelled wheat fiber fractions will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Regular diet with 3 meals a day (minimal 5 times a week)
* BMI between 18.5 and 27 kg/m2

Exclusion Criteria:

* Calorie restricted diet or other special diet during the study or during the last month prior to the study
* Antibiotics in the month prior to the study
* Former surgeries on the gastrointestinal tract, with the exception of an appendectomy
* use of the following types of medications with effects on the gastrointestinal tract during the last 2 weeks prior to the study (spasmolytica, anti-diarrhea, anti-constipation, probiotics)
* Chronic disease of the gastrointestinal tract such as Crohn's disease, ulcerative colitis, irritable bowel syndrome, chronic constipation, chronic frequent diarrhea, clinically relevant lactose intolerance
* Pregnancy, pregnancy desire or breastfeeding
* Diabetes (type 1 and 2)
* Blood donation in the past 3 months prior to the study
* Abnormal hemoglobin (Hb) levels in blood, men must have a Hb level between 14.0 and 18.0 g / dL and women between 12.0 and 16.0 g / dL
* Participation in studies in the past year in which radiation was used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Quantification of acetate, propionate and butyrate production in the colon after consumption of each wheat derived fiber fraction | 2 years